CLINICAL TRIAL: NCT00005750
Title: School and Family-Based Obesity Prevention for Children
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5078; R01HL054102 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2001-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To conduct an integrated, multiple-component, school- and community-based intervention targeting both primary and secondary prevention of obesity among third-fourth-and fifth-graders ("School- and Family-Based Obesity Prevention for Children").

DETAILED DESCRIPTION:
BACKGROUND:

An estimated 25-40 percent of United States pre-adolescents and adolescents are obese. Higher rates have been noted among minority youth. Onset of obesity in late childhood and early adolescence is associated with increased risks of "tracking" of obesity into adulthood, subsequent obesity-related morbidity and mortality, and obesity- related psychosocial morbidity. However, there is limited ability to accurately identify those children who will become obese adults and those who will suffer obesity-related morbidities, Existing treatments for child and adolescent obesity have yielded modest, unsustained effects, and single-component prevention interventions have been relatively ineffective.

DESIGN NARRATIVE:

The intervention model was derived from principles of Bandura's social cognitive theory, and included activities in the school, and the home, and a clinically oriented component for high-risk children. The school component included: a computer-based classroom curriculum; a physical education curriculum; and a school lunch intervention. The home component included correspondence materials and a videotape for parents. Children identified as "high risk" were eligible to enroll in an intensive intervention. In addition, several innovative approaches were included: interventions to influence food preferences and television viewing, interventions promoting health advocacy, and computer-assisted instruction.

An "efficacy trial" evaluated the three-year intervention in a cohort of approximately 1200 3rd graders, in 14 ethnically diverse elementary schools, with follow-up in the 6th grade. 7 schools were randomly assigned to the comprehensive intervention, and 7 schools received an attention-placebo classroom curriculum. Anthropometric measures and assessments of food preferences, cardio-respiratory fitness and self-reported behavior, attitudes and knowledge occurred every six months. Parent interviews occurred annually. Although a careful assessment of effects on parents and the schools was conducted, the crucial question was whether the overall intervention had an impact on student adiposity and behaviors.

The primary objective was to significantly reduce the prevalence of obesity, compared to controls, at the end of the three year intervention. Secondary objectives included maintenance of effects at 6-month follow-up, reducing obesity among high-risk children, improving cardio-respiratory fitness, increasing physical activity, decreasing sedentary activity, reducing the prevalence of unhealthful weight control methods, and improving knowledge, attitudes and perceived self-efficacy regarding the adoption of healthful behaviors. In addition, the investigators identified personal, behavioral and environmental (including family) factors prospectively associated with development of obesity, maintenance of normal weight, weight reduction among overweight children and obesity-related behaviors. Finally, they examined longitudinal changes in height, weight, body mass index (BMI), triceps skin fold thickness, and waist and hip circumferences in girls and boys 8 - 12 years of age, with respect to stages of pubertal development.

ELIGIBILITY:
No eligibility criteria

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1996-04; Study Completion 2001-03

REFERENCES:
- [Background] Robinson TN. Reducing children's television viewing to prevent obesity: a randomized controlled trial. JAMA. 1999 Oct 27;282(16):1561-7. doi: 10.1001/jama.282.16.1561. PMID 10546696
- [Background] Robinson TN. Behavioural treatment of childhood and adolescent obesity. Int J Obes Relat Metab Disord. 1999 Mar;23 Suppl 2:S52-7. doi: 10.1038/sj.ijo.0800860. PMID 10340806
- [Background] Robinson TN. Does television cause childhood obesity? JAMA. 1998 Mar 25;279(12):959-60. doi: 10.1001/jama.279.12.959. No abstract available. PMID 9544774
- [Background] Robinson TN, Saphir MN, Kraemer HC, Varady A, Haydel KF. Effects of reducing television viewing on children's requests for toys: a randomized controlled trial. J Dev Behav Pediatr. 2001 Jun;22(3):179-84. doi: 10.1097/00004703-200106000-00005. PMID 11437193
- [Background] Robinson TN, Kiernan M, Matheson DM, Haydel KF. Is parental control over children's eating associated with childhood obesity? Results from a population-based sample of third graders. Obes Res. 2001 May;9(5):306-12. doi: 10.1038/oby.2000.38. PMID 11346672
- [Background] Robinson TN, Wilde ML, Navracruz LC, Haydel KF, Varady A. Effects of reducing children's television and video game use on aggressive behavior: a randomized controlled trial. Arch Pediatr Adolesc Med. 2001 Jan;155(1):17-23. doi: 10.1001/archpedi.155.1.17. PMID 11177057
- [Background] Robinson TN, Chang JY, Haydel KF, Killen JD. Overweight concerns and body dissatisfaction among third-grade children: the impacts of ethnicity and socioeconomic status. J Pediatr. 2001 Feb;138(2):181-7. doi: 10.1067/mpd.2001.110526. PMID 11174614
- [Background] Robinson TN. The epidemic of pediatric obesity. West J Med. 2000 Oct;173(4):220-1. doi: 10.1136/ewjm.173.4.220. No abstract available. PMID 11017963
- [Background] Erickson SJ, Robinson TN, Haydel KF, Killen JD. Are overweight children unhappy?: Body mass index, depressive symptoms, and overweight concerns in elementary school children. Arch Pediatr Adolesc Med. 2000 Sep;154(9):931-5. doi: 10.1001/archpedi.154.9.931. PMID 10980798